CLINICAL TRIAL: NCT05676554
Title: The Efficacy of a Growth-Mindset Intervention for Adolescents: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk and Suffolk NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETH2223-0067
Record Dates: First submitted 2022-12-20; First posted 2023-01-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Anxiety Disorders and Symptoms; Depression, Anxiety; Adolescent - Emotional Problem
Keywords: Growth Mindset
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will watch the growth mindset session
  Interventions: Other: An Enhanced Psychological Mindset Session for Adolescents
- Waitlist (No Intervention): This arm will receive the intervention once they have completed the follow up at 4 weeks.

INTERVENTIONS:
Other: An Enhanced Psychological Mindset Session for Adolescents — It is a ten-minute psychoeducation video (animation) delivered on the internet, followed by five minutes of stories from fictional students about how they used the concepts. Participants then complete three multiple choice questions aimed to assess their understanding and ability to apply concepts from the video, followed by 'letter of advice' task where participants have to give advice to a fictional younger student based on the information presented in the animation and videos.
  The intervention itself was developed by Perkins et al (2021) based on promoting a growth mindset. It was deemed to be a feasible and acceptable tool to promote mental health (Perkins et al., 2021) in their feasibility trial.
  Arms: Intervention

SUMMARY:
This study is exploring an animated learning resource that could be used online to promote mental health. It is computer based and delivered in a single session, lasting 30 minutes. It teaches young people about thoughts, feelings, personality and the brain, it includes ideas about "mindsets" - or beliefs about the brain - which may be helpful in day-to-day life.

The investigators will use social media to recruit 14-18-year-olds to take part in our research. They will be randomly put into one of two groups - either a group who receive the online session first or a group who receive the session later (at the end of the study).

The animated learning resource aims to promote and protect mental health. The investigators predict it might have some benefits for emotional wellbeing, though the investigators do not know for certain. Young people who take part might learn something new or find it rewarding to know they have been part of research which could be used to help promote mental health.

It is important to know that this is a research study and not a form of treatment for mental health problems.

DETAILED DESCRIPTION:
The study will be advertised on different social media platforms and shared online by the researcher. Participants will be able to click the link for more information where detailed study information will be provided and a link to the study on Qualtrics. The participants will then be able to tick to consent to taking part in the research, then allocated a research identification number which will be linked to their email address.

Once consented demographic information will be collected and baseline measures will be administered (RCADS-11; AFQ-Y8; IPTQ 3 items). Once baseline measures are completed the participants will be randomised by an independent source (via Qualtrics) to either treatment or control (so neither participants or researchers know until after enrolment).

Following randomisation, those who are allocated to the treatment arm will complete 'An Enhanced Psychological Mindset Session for Adolescents' online. A feasibility randomised control trial by Perkins et al. (2021) demonstrated that their enhanced psychological mindset session for adolescents (which is used in this current study) is feasible, acceptable, and potentially scalable. Their single session intervention (SSI) was developed specifically for adolescents and aims to promote emotional wellbeing through encouraging a "growth mindset" as research suggests those with growth mindsets who believe personal traits can change are less likely to experience mental health problems (Schleider et al., 2015).

In total the intervention (watching the video, questions and letter task) takes approximately 30 minutes to complete and the feasibility study took a maximum of 2 hours (including to go through information sheet, consenting process, measures and follow ups). Once the intervention has been completed participants will then be contacted four weeks later for a follow up and asked to complete all measures again. At the end of the trial when all the treatment arm participants have completed the intervention, the control group will be given the link to access it. There will also be a prize draw for those who complete the follow up with a chance to win an amazon voucher (15 £10 vouchers).

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18 years old
* Currently in the United Kingdom

Exclusion Criteria:

* Not currently in the United Kingdom
* Participants who cannot read/write English (by self-selecting to take part in the research they will be able to read English sufficiently to continue),

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
11-item Revised Child Anxiety and Depression Scale (RCADS) (Radez et al., 2021) | Baseline
  Measures anxiety and depression symptoms. It contains six items addressing anxiety symptoms and five addressing depression symptoms, with the option of a two-item impact supplement. It is an 11 item self-report measure using a Likert scale from 0 (Never) to 3 (Always). Higher scores indicate higher reported symptoms with cut off scores provided to indicate clinically significant scores. The measure should take less than five minutes to complete
11-item Revised Child Anxiety and Depression Scale (RCADS) (Radez et al., 2021) | 4 week follow up
  Measures anxiety and depression symptoms

SECONDARY OUTCOMES:
Three items from the Implicit Personality Theory Questionnaire (IPTQ) (Yeager et al., 2013) | Baseline
  Three items from the Implicit Personality Theory Questionnaire (IPTQ) will be used to assess participants views on whether personality is fixed or malleable (Yeager et al., 2013) these items are identical to the ones used in the feasibility study. The self-report three items are: "You have a certain personality, and it is something that you can't do much about," "Your personality is something about you that you can't change very much," and "Either you have a good personality or you don't, and there is really very little you can do about it." The items are rated on a Likert scale from 1 (really disagree) to 6 (really agree), with a higher score suggesting a more fixed mindset. This measure should take less than a few minutes to complete.
Three items from the Implicit Personality Theory Questionnaire (IPTQ) (Yeager et al., 2013) | 4 week follow up
  Used to assess participants views on whether personality is fixed or malleable
The Acceptance and Fusion Questionnaire for Youth-Short Form (AFQ-Y8; Greco et al., 2008) | Baseline
  Used to assess psychological flexibility (being present, aware, and accepting of our thoughts and emotions and acting on values rather than short-term impulses [(Hülsheger et al., 2013]), which captures third-wave cognitive behavioural (e.g., Neff, 2003; Hayes et al., 2011) constructs such as acceptance and values-accordant behaviour. This measure was also used in the feasibility study.
  The AFQ-Y8 is an eight item self-report measure which uses a Likert scale from 0 (not at all true) to 5 (very true). Possible scores range from 0 to 32. There are no clinical cut off scores, but lower total scores indicate greater psychological flexibility.
The Acceptance and Fusion Questionnaire for Youth-Short Form (AFQ-Y8; Greco et al., 2008) | 4 week follow up
  Used to assess psychological flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No